CLINICAL TRIAL: NCT02771431
Title: The Use of Videoconferencing for Monitoring of Patients Post Urologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Manish Vira, Attending Urologist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-659
Record Dates: First submitted 2016-02-22; First posted 2016-05-13 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Urology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): Group 1 will consist of patients receiving in-person attending-patient encounters while inpatients.
- Tele-rounding (Experimental): Group 2 will consist of patients receiving video-conference attending-patient encounters. The intervention is being seen via ipad
  Interventions: Other: Tele-rounding in post operative care

INTERVENTIONS:
Other: Tele-rounding in post operative care — Both groups will receive standard of care. The only difference between these groups would be the physical presence of the attending in the room. Both groups will receive a physical exam with supervision of the attending, one group will have attending in the room and the other will have the attending present via I-pad. In both cases if there was something of concern the attending would step in for the physical exam if needed, regardless of which group they were randomized for.
  Arms: Tele-rounding

SUMMARY:
Our study would be the first randomized study investigating the use of video conferencing via tablet computers versus traditional bedside rounding and its effect on clinical data such as length of stay and complications as well as patient satisfaction. As technology improves, medicine has an obligation to incorporate this technology to improve efficiency and cost-effectiveness. If telerounding is proven to not change outcomes or patient satisfaction, it saves time for the physician during office hours to see more patients or be productive in other ways. Telerounding could be applied in remote areas with a dearth of specialists, allowing these specialists' expertise to reach areas it could not before.

DETAILED DESCRIPTION:
As the healthcare system in America is evolving, doctors are becoming hard-pressed to see and treat more patients in the same amount of time. Over the past century, different forms of "telemedicine" have allowed doctors to treat patients from a distance, in hopes of increasing access to medical care. Several studies have evaluated the utility of telemedicine in the ICU setting, namely using video-conferencing technology to allow ICU attending physicians to monitor their patients with audio and video media more closely. A prospective, step-wedge study by Lily showed that the use of telemedicine reduced adjusted odds mortality and length of stay in the ICU, as well as several complications such as stress ulcers, deep venous thromboses, and ventilator associated pneumonia. Similar conclusions were found by a meta-analysis in 2011 that looked at 176 tele-ICU articles, which included 41,374 patients. With telemedicine technology, intensivists can theoretically have 24-hour oversight of the ICU from a remote location, possibly being able to oversee multiple units.

Although the average urology patient does not require as frequent monitoring as the ICU patient, telemedicine may still play a role in facilitating care for the postoperative urologic patient. In 2004, Ellison el al conducted a study comparing patient satisfaction between patients seen via standard bedside rounds, patients seen via telerounds (as an additional visit) through a laptop computer, and patients only seen via telerounds through a remotely controlled robot. This study showed that telerounding (either of the latter two arms) was associated with greater patient satisfaction in postoperative care, which was found to be linked to physician availability4. In 2007, the same authors conducted a randomized study investigating morbidity, length of stay, and patient satisfaction between standard bedside rounds versus robotic telerounding. There were no differences in outcomes between the two groups. A significant limitation of robotic telerounding is cost. Having and maintaining the robot costs around $60,000 per year, although Gandas et al was able to find a positive financial impact when using the robot in postoperative gastric bypass patients6. However, the development of tablet computers, which have user-friendly video-conferencing applications, has made telemedicine a more affordable tool. In 2012, Kacsmarek et al conducted the first study using tablet computers investigating post-operative patient satisfaction. Their study demonstrated that tablet telerounding can significantly enhance patients' post-operative experience by providing quicker face-to-face access with their attending physician.

Our study would be the first randomized study investigating the use of video conferencing via tablet computers versus traditional bedside rounding and its effect on clinical data such as length of stay and complications as well as patient satisfaction. As technology improves, medicine has an obligation to incorporate this technology to improve efficiency and cost-effectiveness. If telerounding is proven to not change outcomes or patient satisfaction, it saves time for the physician during office hours to see more patients or be productive in other ways. Telerounding could be applied in remote areas with a dearth of specialists, allowing these specialists' expertise to reach areas it could not before.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Undergo elective Urologic surgery requiring post-operative inpatient stay

Exclusion Criteria:

1. Patients under 18 years of age
2. Patients who are unable to provide their own consent
3. Patients who undergo urgent or emergent Urologic procedures who are not already enrolled in the study
4. Patients who do not require an inpatient post-operative stay
5. Patients who are seen on the weekend (Saturday or Sunday)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Complication rates | 4 years
length of inpatient stay | 4 years
number of lab tests ordered | 4 years
severity of complications | 4 years

SECONDARY OUTCOMES:
Additionally patient satisfaction will be looked at based on post-operative questionnaire. | 4 years
  how satisfied they were with seeing provider remotely vs standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Manish Vira, MD, Principal Investigator — Physician
Locations (1):
- North Shore LIJ, New Hyde Park, New York, United States

REFERENCES:
- [Background] Strehle EM, Shabde N. One hundred years of telemedicine: does this new technology have a place in paediatrics? Arch Dis Child. 2006 Dec;91(12):956-9. doi: 10.1136/adc.2006.099622. PMID 17119071
- [Background] Lilly CM, Cody S, Zhao H, Landry K, Baker SP, McIlwaine J, Chandler MW, Irwin RS; University of Massachusetts Memorial Critical Care Operations Group. Hospital mortality, length of stay, and preventable complications among critically ill patients before and after tele-ICU reengineering of critical care processes. JAMA. 2011 Jun 1;305(21):2175-83. doi: 10.1001/jama.2011.697. Epub 2011 May 16. PMID 21576622
- [Background] Young LB, Chan PS, Lu X, Nallamothu BK, Sasson C, Cram PM. Impact of telemedicine intensive care unit coverage on patient outcomes: a systematic review and meta-analysis. Arch Intern Med. 2011 Mar 28;171(6):498-506. doi: 10.1001/archinternmed.2011.61. PMID 21444842
- [Background] Ellison LM, Pinto PA, Kim F, Ong AM, Patriciu A, Stoianovici D, Rubin H, Jarrett T, Kavoussi LR. Telerounding and patient satisfaction after surgery. J Am Coll Surg. 2004 Oct;199(4):523-30. doi: 10.1016/j.jamcollsurg.2004.06.022. PMID 15454133
- [Background] Ellison LM, Nguyen M, Fabrizio MD, Soh A, Permpongkosol S, Kavoussi LR. Postoperative robotic telerounding: a multicenter randomized assessment of patient outcomes and satisfaction. Arch Surg. 2007 Dec;142(12):1177-81; discussion 1181. doi: 10.1001/archsurg.142.12.1177. PMID 18086984
- [Background] Gandsas A, Parekh M, Bleech MM, Tong DA. Robotic telepresence: profit analysis in reducing length of stay after laparoscopic gastric bypass. J Am Coll Surg. 2007 Jul;205(1):72-7. doi: 10.1016/j.jamcollsurg.2007.01.070. PMID 17617335
- [Background] Kaczmarek BF, Trinh QD, Menon M, Rogers CG. Tablet telerounding. Urology. 2012 Dec;80(6):1383-8. doi: 10.1016/j.urology.2012.06.060. PMID 23206790